CLINICAL TRIAL: NCT00105976
Title: A Phase 2, Double-Blind, Parallel, Placebo-Controlled, Randomized Study to Evaluate the Efficacy and Safety of 3 Different Dose Levels (2.5, 7.5 and 20 mg) of MM-093 in Patients With Active Rheumatoid Arthritis on Stable Doses of Methotrexate
Brief Title: Efficacy Study of MM-093 in Rheumatoid Arthritis Patients on Methotrexate (MTX)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MM-093-01-200
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

INTERVENTIONS:
Drug: MM-093

SUMMARY:
The purpose of this clinical study is to see if an experimental drug, called MM-093, is safe and effective in the treatment of rheumatoid arthritis. MM-093 is a genetically engineered version of a naturally occurring protein called alpha fetoprotein (AFP). Adults normally have very small amounts of AFP in their bloodstream. However, during pregnancy, AFP levels in both the mother and the fetus are much higher than normal. It has been observed that women with RA (Rheumatoid Arthritis) have fewer symptoms during pregnancy, particularly during the third trimester. At this time, the levels of AFP in the blood of the mother and fetus are the highest. This observation led researchers to begin examining AFP as a possible treatment for RA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* Meet ACR (American College of Rheumatology) criteria for RA
* Have active RA consisting of 6 or more swollen and 6 or more tender joints
* Have RA for at least 6 months
* Had disease onset after 16 years old
* Currently being treated with a stable, well-tolerated dose of MTX (10 to 25 mg) given once weekly for at least 6 consecutive weeks prior to the screening visit
* Currently being treated with folic acid
* Willing to remain on a constant, once-weekly dose of MTX and folic/folinic acid throughout the duration of the study.
* Understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures being performed.
* Be able and willing to comply with study visits and procedures per protocol.
* Sexually active men must agree to use a medically acceptable form of contraception during the study and continue for 4 weeks after the last dose of study drug.
* Women of childbearing potential must use a medically acceptable means of birth control during the study and for 4 weeks after the last dose
* Must be able to store study drug in a refrigerator at home

Exclusion Criteria:

* Use of any B-cell depleting therapy in the last 6 months
* Use of Leflunomide or Humira in the last 3 months
* Use of any investigational drug or biologic agent in the last 2 months
* Use of Remicade in the last 2 months
* Use of cyclosporine, sulphasalazine, auranofin, intramuscular gold, azathioprine, D-penicillamine or tacrolimus within the last 6 weeks
* Use of more than 10 mg/day of prednisone or equivalent in the last 4 weeks
* Use of intra-articular corticosteroid injection in the last 4 weeks
* Use of a bolus IM/IV (intramuscular/intravenous) treatment with corticosteroids (>20 mg prednisone or equivalent) in the last 4 weeks
* Use of Enbrel in the last 4 weeks
* Use of Kineret in the last 2 weeks
* Current use of more than 1 NSAID (non-steroidal anti-inflammatory drug) or dose of NSAID greater than the maximum recommended dose in the product information
* Cancer, or a history of cancer (other than successfully resected cutaneous basal and squamous cell carcinoma) within 5 years before the screening visit.
* Any condition for which participation in this study is judged by the physician to be detrimental to the patient, such as history of significant or unstable cardiac, pulmonary, gastrointestinal, neurological, or psychiatric disease, or a DMARD (Disease-Modifying Anti-Rheumatic Drug)-related severe, potentially life-threatening AE (Adverse Event).
* Significant ongoing infection requiring systemic antibiotic, antifungal, antiviral, or any anti-mycobacterial therapy.
* Autoimmune or connective tissue disorder other than rheumatoid arthritis (e.g. systemic lupus erythematosis, scleroderma or psoriatic arthritis).
* Grade 2 or above leukopenia (i.e. white blood cells < 3000/mm3 [SI units: < 3.0 x 10^9/L]).
* Thrombocytopenia or thrombocytosis (platelets < 125,000/mm3 or ≥ 1,000,000/mm3 [SI units: < 125 x 10^9/L or ≥ 1,000 x 10^9/L]), respectively.
* Grade 2 or above liver function abnormality (i.e. total bilirubin > 1.5 x the upper limit of normal; or aspartate aminotransferase [AST/SGOT] or alanine aminotransferase [ALT/SGPT] > 2.5 x upper limit of normal).
* Renal disease (including serum creatinine level > 1.5 x the upper limit of normal).
* Any history of immunodeficiency syndromes or infection with human immunodeficiency virus (HIV), or a history of hepatitis C or chronic hepatitis B.
* Pregnant or breastfeeding women or women planning to become pregnant during the study or within 4 weeks after the last dose of study drug.
* Any major surgery, including joint surgery, within 3 months before screening visit.
* Scheduled elective surgery during study participation.
* Participated in any previous clinical trial using MM-093 or have any prior exposure to MM-093.
* History of severe hypersensitivity to goat, sheep or cow milk or products derived from goat, sheep or cow milk (patients who are lactose intolerant are not excluded).
* Any other condition that the investigator feels would jeopardize the integrity of the study (e.g. a CTCAE [Common Terminology Criteria for Adverse Events] grade 2 or above clinical finding or laboratory result).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2005-02

PRIMARY OUTCOMES:
To evaluate the efficacy of 3 different dose levels of MM-093 as measured by the percentage of patients achieving an ACR20 response after 24 weeks compared to placebo
To evaluate the safety and tolerability of 3 different dose levels of MM-093

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - University of Alabama, Birmingham, Alabama
  - Montgomery Rheumatology Associates, Montgomery, Alabama
  - Arizona Arthritis Research, PLC, Paradise Valley, Arizona
  - ArthroCare, Arthritis Care and Research, Inc., Phoenix, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Arthritis Medical Center of the Central Coast, Santa Maria, California
  - Boling Clinical Trials, Upland, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - New England Research Associates, Bridgeport, Connecticut
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Renstar Medical Research, Ocala, Florida
  - International Medical Research, Ormond Beach, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Center for Arthritis and Rheumatic Diseases, South Miami, Florida
  - Coeur d'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Illinois Bone and Joint Institute, Morton Grove, Illinois
  - The Arthritis Center, Springfield, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Rheumatology Associates, PC, Indianapolis, Indiana
  - Wichita Clinic, Wichita, Kansas
  - Rx Trials, Inc., Columbia, Maryland
  - Arthritis Center of Nebraska, Lincoln, Nebraska
  - Arthritis Center of Reno, Reno, Nevada
  - Arthritis, Osteoporosis & Musculoskeletal Disease Center, Concord, New Hampshire
  - Arthritis Health Associates, Syracuse, New York
  - Asheville Rheumatology and Osteoporosis Research Associates, Inc, Asheville, North Carolina
  - Arthritis Clinic and Carolina Bone and Joint PA, Charlotte, North Carolina
  - CARE Center, Raleigh, North Carolina
  - North Carolina Arthritis and Allergy Care Center, Raleigh, North Carolina
  - Veterans Administration Research Services, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - The Arthritis Group, Memphis, Tennessee
  - Austin Rheumatology Research, Austin, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Arthritis and Osteoporosis Clinic, Waco, Texas
  - University of Utah Division of Rheumatology, Salt Lake City, Utah